CLINICAL TRIAL: NCT03504293
Title: Sahlgrenska EUS ERCP Study
Brief Title: The Diagnostic Value of Combinatory EUS and ERCP in Unclear Lesions
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Per Hedenström, MD PhD, Sahlgrenska University Hospital
Other Study IDs: EUS-ERCP Study
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Neoplasms; Biliary Stricture; Biliary Tract Neoplasms; Biliary Tract Diseases
Keywords: Endosonography; Endoscopic retrograde choledochography
MeSH Terms: conditions — Neoplasms; Biliary Tract Neoplasms; Biliary Tract Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Combinatory EUS and ERCP — EUS performed as a supplementary procedure in addition to ERCP

SUMMARY:
ERCP with brush cytology has a poor to moderate accuracy in unclear biliary lesions. Endoscopic ultrasound (EUS) with fine needle aspiration (FNA) for cytology may override some of these shortcomings.

The current prospective study, performed in a tertiary University center, aims to study the feasibility, the accuracy and the clinical value of combinatory ERCP and EUS in unclear biliary lesions.

DETAILED DESCRIPTION:
The eligible study participants with unclear biliary lesions referred for an ERCP to the Sahlgrenska Univeristy Hospital endoscopy unit will be subjected to ERCP with/without brush cytology followed by EUS with/without FNA.

The results of ERCP and EUS will be compared to the pathology report of surgical specimens in resected patients or to clinical follow up at 12 months post-EUS in non-resected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unclear lesions or strictures in the biliary tract referred for endoscopy work up

Exclusion Criteria:

* Patients unwilling to participate
* Patients unfit for EUS and ERCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unclear lesions or strictures in the biliary tract
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 12 months post-EUS
  Overall accuracy of ERCP and EUS

SECONDARY OUTCOMES:
Adverse event rate | 30 days post-EUS
  The number of patients ending up with some type of complication related to ERCP or EUS

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Sadik, Ass Prof, Principal Investigator — Sahlgrenska University Hospital, Gothenburg
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No